CLINICAL TRIAL: NCT01342991
Title: Randomised Controlled Trial of Open Milligan-Morgan Haemorrhoidectomy Versus Laser Closed Haemorrhoidectomy
Brief Title: Trial of Open Milligan-Morgan Haemorrhoidectomy Versus Laser Closed Haemorrhoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Lincolnshire and Goole Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mr PJ Moore, Consultant Surgeon, Northern Lincolnshire and Goole Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09/H1305/59
Record Dates: First submitted 2011-04-14; First posted 2011-04-27 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Haemorrhoids; Haemorrhoidectomy; Milligan-Morgan Haemorrhoidectomy; Open Haemorrhoidectomy
Keywords: Haemorrhoids; Haemorrhoidectomy; Laser Haemorrhoidectomy; Milligan-Morgan Haemorrhoidectomy; Open Haemorrhoidectomy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milligan-Morgan Haemorrhoidectomy (Active Comparator): Control arm
  Interventions: Procedure: Laser Haemorrhoidectomy
- Laser Haemorrhoidectomy (Experimental): This new method of haemorrhoidectomy is being compared to the standard Milligan-Morgan Haemorrhoidectomy.
  Interventions: Procedure: Laser Haemorrhoidectomy

INTERVENTIONS:
Procedure: Laser Haemorrhoidectomy — The intervention comprises laser haemorrhoidectomy
  This procedure will be performed under local anaesthetic with sedation as a day case
  The haemorrhoids are excised using sharp dissection (over a clamp) and the cut edges are sealed using CO2 laser.
  Pre-operative local anaesthesia will be given
  Other Names: Laser Seal Haemorrhoidectomy
  Arms: Milligan-Morgan Haemorrhoidectomy
Procedure: Laser Haemorrhoidectomy — The intervention comprises laser haemorrhoidectomy
  This procedure will be performed under local anaesthetic with sedation as a day case
  The haemorrhoids are excised using sharp dissection (over a clamp) and the cut edges are sealed using CO2 laser.
  Pre-operative local anaesthesia will be given
  Arms: Laser Haemorrhoidectomy

SUMMARY:
This is a randomised trial to compare both the procedures and the difference in their immediate postoperative pain, recovery and quality of life.

DETAILED DESCRIPTION:
Haemorrhoidectomy (excision of haemorrhoids) is the procedure of choice for grade 3 & 4 symptomatic haemorrhoids. The standard technique in the UK (open Milligan-Morgan) is to excise the haemorrhoids under general anaesthetic (typically using electrocautery) leaving raw areas in anal canal. As a result, patients often experience significant post operative pain which can impact on patient function for weeks following surgery. This would be considered as the gold standard for the operative treatment for haemorrhoids. Due to the difficult post operative recovery of this procedure, alternative techniques for performing haemorrhoidectomy have been explored. One approach, which is gaining some popularity, is stapled haemorrhoidectomy [1]. In this technique, a circular stapling device is used to excise proximal mucosa in order to disconnect the haemorrhoidal blood supply and to pull up the haemorrhoidal mass. The edges of the excised mucosa are simultaneously closed with a row of staples. In a recent meta-analysis of 29 randomised controlled trials including 2056 patients, stapled haemorrhoidectomy was associated with reduced postoperative pain and reduction in return to activity by nearly 12 days in comparison to open haemorrhoidectomy [2]. Although postoperative complication rates were similar, stapled haemorrhoidectomy was associated with significantly more recurrences in the longer term (relative risk 2.29). The stapled haemorrhoidectomy technique has not gained universal acceptance. This may be related to the cost and availability of stapling devices in many centres.

Unlike specialized stapling devices, lasers are widely available in the operating theatre and are used in many operations to cauterise tissue. The resulting burn is superficial in comparison to electrocautery. Consequently, lasers have been used to perform open haemorrhoidectomy with the expectation of reducing post operative pain. However, randomised trials comparing the use of lasers versus cold scalpel for open haemorrhoidectomy have shown no significant differences in post operative pain [3]. Although, the laser appears to offer no advantage in open haemorrhoidal procedures, an alternative technique for laser haemorrhoidectomy has been developed by Peter Thompson from Laser Haemorrhoid Centre in Phoenix, Arizona. In this alternative technique, a laser is used to seal the raw mucosal edges after excision of the piles. In common with stapled haemorrhoidectomy, the mucosa is sealed closed rather than left open. Consequently, patients appear to experience markedly less post operative pain. The technique is also simple and quick with a shallow learning curve. Due to the speed and relative comfort of the procedure, patients may be routinely operated on using sedation and local anaesthetic, rather than full general anaesthetic which is standard practice for most haemorrhoidectomies.

Over the last 2 years,the investigators have performed laser haemorrhoidectomy for 60 patients. The age range was 32 to 81 years .The ratio for male: female was 31:29. All were done under local anaesthesia with sedation except one (1.6%) which was converted to general anaesthesia. All patients except 2 (3.5%) were discharged within two hours of operation. One was delayed due to administration of general anaesthesia and the second one was admitted for post operative bleeding and was actively observed for three days, after which he was discharged. There were four re-admissions (6.6%), two had post operative oedema & two had oedema and pain. All of them were actively observed and discharged later. Four patients (6.6%) also developed chronic anal fissures post operatively, two of them healed with six weeks course of Glyceryl Tri Nitrate (GTN) cream and the other two are on conservative management for non-healing fissures.

The investigators wish to objectively determine whether laser closed haemorrhoidectomy is associated with significantly less post operative pain and an earlier return to function in comparison to the Milligan-Morgan Haemorrhoidectomy which is the standard procedure performed across the trust.

ELIGIBILITY:
Inclusion Criteria:

* Are fit enough to undergo general anaesthesia
* Are between the age of 18 and 80 years
* Are able and willing to provide informed consent
* Show no preference to either operative procedure and agree to randomization
* No contra-indications to receiving laser treatment

Exclusion Criteria:

* Are not fit enough to undergo a general anaesthesia
* Are not over the age of 18 years
* Are unable or unwilling to provide informed consent
* Have stated their operation preference
* Have any contra-indication preventing them from receiving laser treatment
* Have a history of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Post operative pain relief | 6 weeks post-operatively
  Visual Analogue Score (1 to 10) willbe used to quantitatively assess pain outcomes.

SECONDARY OUTCOMES:
Quality of life | Immediately pre-operatively and again at 6 weeks post-operatively
  SF12 forms will be filled by the patients pre-operatively and again at 6 weeks post-operatively to assess any change in the quality of life this procedure may provide and compare the results between the two procedures.
analgesia consumption | 6 weeks post-operatively
  patients maintain a pain medication diary in which they document the amount of analgesia they have consumed in the post-operative period.
  They are all given a standard regime of analgesics post-operatively unless there are any contra-indications.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Moore, MD, FRCS, Principal Investigator — Northern Lincolnshire and Goole Hospitals NHS Foundation Trust
Locations (1):
- Northern Linconshire & Goole NHS Foundation trust, Goole, North Lincolnshire, United Kingdom